CLINICAL TRIAL: NCT02592187
Title: A Cognitive Training Tool Based on Life-logging in Mild Cognitive Impairment (ReMemory-MCI)
Acronym: ReMemory-MCI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Consorci Sanitari de Terrassa (Other)
Collaborators: University of Barcelona (Other); Associació Vallès Amics de la Neurologia (Other); Fundació La Marató de TV3 (Other)
Responsible Party: Principal Investigator, Maite Garolera, Doctor, Consorci Sanitari de Terrassa
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Fundacio la MaratóTV3 20141510
Record Dates: First submitted 2015-07-31; First posted 2015-10-30 (Estimated); Last update posted 2019-01-11 (Actual); Status verified 2019-01

CONDITIONS: Mild Cognitive Impairment
Keywords: Life-logging; Cognitive Training; Mild Cognitive Impairment; Memory; Information and communications technology (ICT) in healthcare; Portable camera
MeSH Terms: conditions — Cognitive Dysfunction

ARMS (2):
- Experimental intervention (Experimental): ReMemory-MCI training
  Interventions: Behavioral: ReMemory-MCI training
- Control intervention (Active Comparator): Control intervention
  Interventions: Behavioral: Control intervention

INTERVENTIONS:
Behavioral: ReMemory-MCI training
  Arms: Experimental intervention
Behavioral: Control intervention
  Arms: Control intervention

SUMMARY:
Background: Mild Cognitive Impairment (MCI) is a risk factor for dementia and represents a critical window of opportunity to intervene and alter the trajectory of both cognitive and functional decline. Emerging life-logging technologies has shown a tremendous potential to increase autobiographical memory.

Objective: The main goal of the present study is to develop a Cognitive Training program (CT) for MCI based on life-logging captured by a Wearable Camera (WeC) recording specific autobiographical episodes for stimulating posteriorly episodic memory. The challenge is to create an application to manage this large collection of images, which can be easily retrieved as events by users in a therapeutic context as a multimodal cognitive stimulation. The investigators will conduct a quasi-experimental design with non-equivalent control group, evaluating the effectiveness of the life-logging re-experiencing program immediately and 3-month follow-up period.

Methodology: The design is a pretest, posttest and follow-up design, where 30 adults with MCI were sequentially allocated to one of two conditions: intervention or control group. All subjects wore a lifelogging WeC during two weeks, and subsequently they were generated several videos with the most relevant information of each event. Subjects in the Intervention Group will attend 1-hour individual training sessions 2 times per week for 14 8 weeks. Main outcomes measures will be cognitive, functional, emotional and quality of life measures, as well as biochemical measures (BDNF).

Expected results: The investigators expect the outcomes to provide preliminary evidence that autobiographical experimentation CT programs can positively impact cognitive functioning and may represent an effective strategy to improve memory and functionality in those who begun to experience cognitive decline.

ELIGIBILITY:
Inclusion Criteria:

* 65-90 years of age
* Meet definition criteria for MCI (Petersen, 2004)
* Be receiving CT at least three month in Day Hospital during three months or more; c) having memory complaint, usually verified by an informant
* Having memory complaint, usually verified by an informant
* Memory performance below the mean score for the corresponding age and education group
* Having normal general cognitive functioning as determined by a Mini-Mental State Examination (MMSE) score > o = 24
* Having a reliable caregiver who can supervise the patient's daily activities
* Having Global clinical dementia rating scale score of 0.5
* Granted written informed consent accepting to participate in the study

Exclusion Criteria:

* Neurological, psychiatric or unstable medical disorders
* Intellectual deficiency (Premorbid Intellectual Quotient (IQ) -Vocabulary- less 85)
* Relevant hearing, vision, motor or language deficits
* Less than 4 years of education e) acquisition of Catalonian or Spanish languages after 15 years old

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-06; Primary Completion 2019-02 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
Change in memory after receiving treatment | after 16 sessions treatment and 3 months
  Memory was measured using the Logical Memory Test from the Wechsler Memory Scale, IV version (WMS-IV, Spanish version); the International Shopping List Task and the One Card Learning Task from the computerized neurocognitive battery Cogstate.
Change in attention after receiving treatment | after 16 sessions treatment and 3 months
  Attention was measured using the Identification Task from the computerized neurocognitive battery Cogstate and the Forward Digit Span from the Wechsler Adult Intelligence Scale, fourth edition (WAIS-IV)
Change in working memory after receiving treatment | after 16 sessions treatment and 3 months
  orking memory was measured using the One Back Task from the computerized neurocognitive battery Cogstate and the Backward Digit Span from the Wechsler Adult Intelligence Scale, fourth edition (WAIS-IV).
Change in executive function, set-shifting after receiving treatment | after 16 sessions treatment and 3 months
  Set-shifting was measured using the Colors Trails Test
Change in executive function,verbal fluency | after 16 sessions treatment and 3 months
  erbal Fluency was measured using the Controlled Oral Word Association Test, spanish adaptation, and semantic fluency test using the category Animals
Change in executive function, inhibition after receiving treatment | after 16 sessions treatment and 3 months
  Inhibition was measured using the Five Digit Test
Change in processing speed after receiving treatment | after 16 sessions treatment and 3 months
  Processing speed was measured using the Detection Task from the computerized neurocognitive battery Cogstate battery

SECONDARY OUTCOMES:
Change in subjective memory complaints after receiving treatment | after 16 sessions treatment and 3 months
  subjective memory complaints was measured using Memory Faiures of EveryDay (MFE) Test
Change in functional capacity after receiving treatment | after 16 sessions treatment and 3 months
  Functional capacity was measured using Functional Assessment Questionnaire (FAQ) and the UCSD Performance-Based Skills Assessment (UPSA).
Change in depression and anxiety after receiving treatment | after 16 sessions treatment and 3 months
  depression and anxiety were measured using the Hospital Anxiety and Depression Scale (HADS)
Change in quality of life | after 16 sessions treatment and 3 months
  Quality of life was measured using Quality of Life-Alzheimer Disease (QoL-AD)
Change in Neuropsychiatric symptoms | after 16 sessions treatment and 3 months
  Neuropsychiatric symptoms was measured using Neuropsychiatric Inventory Questionnaire (NPI)
Change in Caregiver Burden | after 16 sessions treatment and 3 months
  Caregiver Burden was measured using the Zarit Caregiver Burden Scale
Change in patient's self-esteem | after 16 sessions treatment and 3 months
  Self-Esteem was measured using the Rosenberg Self-Esteem Scale
Change in patient and caregiver's perception of social support | after 16 sessions treatment and 3 months
  Perception of social support was measured using the Duke-UNC Functional Social Support Questionnaire
Change in neuroplasticiy | after 16 sessions treatment and 3 months
  neuroplasticiy was measured using Brain-derived neutrophic factor (BDNF) serum levels

CONTACTS AND LOCATIONS:
Overall Officials: Maite Garolera, PhD, Principal Investigator — Consorci Sanitari de Terrassa